CLINICAL TRIAL: NCT00476216
Title: Phase I Feasibility Study of the Combination of Fondaparinux (Arixtra) With Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Fondaparinux (Arixtra) With Chemotherapy for Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor of Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F070309006; UAB 0649 (Other: Institutional study protocol number)
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Non-Small Cell Lung Cancer; Venous Thromboembolism
Keywords: Non-Small Cell Lung Cancer; Venous Thromboembolism; VTE; Arixtra
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Venous Thromboembolism | interventions — Drug Therapy; Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of Arixtra with chemotherapy (Experimental): Carboplatin 6 AUC q 21 days; Paclitaxel 200 mg/m2 q 21 days. Cohort I: Arixtra 2.5 mg SQ qd x 21 days; Cohort II: Arixtra weight-based dose (D1-2)followed by Arixtra 2.5 SQ q day (D3-21)
  Interventions: Drug: Combination of Arixtra with chemotherapy

INTERVENTIONS:
Drug: Combination of Arixtra with chemotherapy — Single arm, 2 cohort feasibility study:
  Carboplatin will be administered intravenously over approximately 30 minutes after paclitaxel infusion is completed and the dose will be calculated on basis of an area under the curve (AUC) of 6, according to the formula administered every 21 days. Paclitaxel will be administered 200 mg/m2 over 3 hours every 21 days.
  Patients in both cohorts 1 & 2 will receive standard chemotherapy alone during cycle 1.
  Cohort 1:During subsequent cycles (2-4) patients will receive a daily prophylactic dose (day 1 through 21) of Arixtra and continue 21 days after the last course of chemotherapy.
  Cohort 2: Patients in cohort 2 will receive standard chemotherapy alone during cycle 1. During subsequent cycles, the patient will receive a therapeutic weight based dose of Arixtra for the first 2 days of each chemotherapy cycle followed by a daily prophylactic dose of Arixtra (day 3 through 21) until the next course of chemotherapy.
  Other Names: Fondaparinux

SUMMARY:
There is a direct association between cancer and thrombosis (blood clots). The purpose of this study is to determine the best dose of an antithrombotic (prevents blood clots) agent called fondaparinux in non-small cell lung cancer(NSCLC). Patients will also receive chemotherapy.

DETAILED DESCRIPTION:
This is a single center, open-labeled, single arm phase 1 feasibility study in patients with newly diagnosed stage IV NSCLC. To evaluate the change in the biologic parameters measured, two cohorts of patients will receive altered dosing regimens of fondaparinux starting with the second cycle of chemotherapy. The biologic parameters measured during the first cycle of chemotherapy will serve as a control for each patient. Chemotherapy consists of 3-week cycles of carboplatin and paclitaxel. The absolute maximum length of therapy with fondaparinux will be 3 months, regardless of which cohort the patient is assigned.

This study consists of 2 cohorts:

Cohort 1:

Patients in cohort 1 will receive standard chemotherapy alone during cycle 1. During subsequent cycles (2-4) patients will receive a daily prophylactic dose (day 1 through 21) of fondaparinux. The anticoagulation will continue 21 days after the last course of chemotherapy.

Cohort 2:

Patients in cohort 2 will receive standard chemotherapy alone during cycle 1. During subsequent cycles, the patient will receive a therapeutic weight based dose of fondaparinux for the first 2 days of each chemotherapy cycle followed by a daily prophylactic dose of fondaparinux (day 3 through 21) until the next course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of Non-Small Cell Lung Cancer.
* Stage IV Non-Small Cell Lung Cancer.
* Measurable or assessable tumor parameters according to RECIST criteria.
* ECOG Performance Status 0-2.
* Age between 18 and 79 years (in the State of Alabama > 18).
* Adequate hematologic, coagulation, liver and renal function, defined as:
* Absolute neutrophil count (ANC) ≥ 1500/µL
* Platelet count ≥ 100,000/µL
* Serum Glutamic Oxaloacetic Transaminase(SGOT)/Serum Glutamic Pyruvic Transaminase(SGPT) ≤ 2.5 x upper limit of normal or ≤ 5 x upper limit of normal when liver metastases are present
* Total bilirubin value ≤ 1.5 x upper limit of normal
* Serum creatinine value ≤ 1.5 x upper limit of normal
* Normal prothrombin time and partial thromboplastin time
* Fully recovered from any previous surgery (at least 4 weeks since major surgery).
* Must have recovered from prior radiation therapy (at least 3 weeks).
* All participants must agree to practice approved methods of birth control (if applicable). A negative pregnancy test must be documented during the screening period for women of childbearing potential.
* Must provide written informed consent and authorization to use and disclose health information.
* No prior chemotherapy.

Exclusion Criteria:

* Active bleeding disorder.
* Evidence of hemoptysis. Patients with blood-tinged or blood-streaked sputum will be permitted on study if the hemoptysis amounts to less than 5 mL of blood per episode and less than 10 mL of blood per 24-hour period in the best estimate of the investigator.
* Previous history of Venous Thromboembolism (VTE) within 12 months and requiring active anticoagulation therapy.
* Concurrent cancer chemotherapy, biologic therapy or radiotherapy.
* Administration of any investigational drug within 28 days prior to administration of the current therapy.
* Symptomatic brain metastases; those patients should be treated first with either whole brain radiation therapy or radiosurgery and have stable disease.
* Concurrent serious infection.
* Concomitant severe or uncontrolled underlying medical disease unrelated to the tumor, which is likely to compromise patient safety and affect the outcome of the study.
* History of other malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for a minimum of 2 years.
* Any evidence or history of hypersensitivity or other contraindications for the drugs used in this trial.
* Psychiatric disorder that prevents patients from providing informed consent or following protocol instructions.
* Pregnant or lactating women.
* Creatinine clearance < 30 mL/min.
* Patient body weight < 50 kg.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The tolerability and safety of the combination of fondaparinux with standard chemotherapy (carboplatin/paclitaxel). | Every 3 weeks prior to each cycle of therapy.

SECONDARY OUTCOMES:
Clinically evident Venous Thromboembolism (VTE) | Every 3 weeks prior to each cyle of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States